CLINICAL TRIAL: NCT03569618
Title: Effect of a Digital Therapeutic on Processing Speed in Adults With Multiple Sclerosis
Brief Title: Digital Cognition in Multiple Sclerosis
Acronym: DigCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-19891
Record Dates: First submitted 2018-03-13; First posted 2018-06-26 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis; Cognitive Decline
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study assessment administrator is blinded to what digital tool the subject has been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Game 1 (Active Comparator): Tablet-based Game 1.
  Interventions: Device: Tablet-based Game
- Game 2 (Placebo Comparator): Tablet-based Game 2.
  Interventions: Device: Tablet-based Game

INTERVENTIONS:
Device: Tablet-based Game — Tablet-based game aimed at improving processing speed and attention.

SUMMARY:
A DIGITAL THERAPEUTIC TO IMPROVE THINKING IN MULTIPLE SCLEROSIS

WHO: 65 participants with a confirmed diagnosis of Multiple Sclerosis (MS)

WHY: Purpose of the study is to compare the effect of 2 tablet-based brain training digital tools on important components of thinking (cognition).

WHAT: Complete a set of tests (physical and cognitive) at baseline, 6 weeks and 14 weeks, and use one of two brain training tools on an iPad in your home, for 25 minutes a day, 5 days a week, for 6 weeks.

WHERE: UCSF WEILL INSTITUTE FOR NEUROSCIENCES (675 Nelson Rising Lane, San Francisco, CA)

DETAILED DESCRIPTION:
The purpose of this study is to begin to test a brain training video game in people with Multiple Sclerosis (MS).

Visit 1. After informed consent, you will complete a series of questions about your functioning and mood. You will then complete a series of tests (vision, hand tapping, walking). Then, you will complete a set of thinking tests. The first set will be paper and pencil. The second set will be on a tablet or a computer. You will use your study code to sign into these tools and you won't provide any personal details for the digitized tests.

Finally, you will complete the "cognitive training tool". There are two versions of this digital, iPad based tool, which takes about 25 minutes to complete and is designed to be entertaining. You will be randomized into 1 of 2 groups: each group will play a version of the brain training game. You will not be told what group/game type you were randomized into. You will be given the tablet with the game on it to take home, and to practice this game 5 times a week for 6 weeks.

Visit 2. After the 6 weeks of at-home training, you will then come back to the research study unit to do a repeat of the initial visit (with physical and cognitive assessments). At this study visit, you will also be returning the iPad.

Visit 3. You will then return 8 weeks after Visit 2, to do a repeat of the assessments.

You will be compensated for each study visit (visit 1: $50, visit 2: $100, visit 3: $150).

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women diagnosed with multiple sclerosis (MS) or clinically isolated syndrome (CIS)
* SDMT z-score range (-2 to +1)
* Wifi available in home
* Able to use a tablet (iPad)
* Able to attend 3 study visits in person.

Exclusion Criteria:

* Clinician's assessment of visual, cognitive, or motor impairment that would preclude participation.
* A clinical relapse within the last 30 days.
* Steroid treatment for clinical relapse within the last 30 days.

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riley Bove, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bove R, Rowles W, Zhao C, Anderson A, Friedman S, Langdon D, Alexander A, Sacco S, Henry R, Gazzaley A, Feinstein A, Anguera JA. A novel in-home digital treatment to improve processing speed in people with multiple sclerosis: A pilot study. Mult Scler. 2021 Apr;27(5):778-789. doi: 10.1177/1352458520930371. Epub 2020 Jun 25. PMID 32584155
- [Derived] Hsu WY, Rowles W, Anguera JA, Anderson A, Younger JW, Friedman S, Gazzaley A, Bove R. Assessing Cognitive Function in Multiple Sclerosis With Digital Tools: Observational Study. J Med Internet Res. 2021 Dec 30;23(12):e25748. doi: 10.2196/25748. PMID 34967751
- [Derived] Hsu WY, Rowles W, Anguera JA, Zhao C, Anderson A, Alexander A, Sacco S, Henry R, Gazzaley A, Bove R. Application of an Adaptive, Digital, Game-Based Approach for Cognitive Assessment in Multiple Sclerosis: Observational Study. J Med Internet Res. 2021 Jan 20;23(1):e24356. doi: 10.2196/24356. PMID 33470940

RESULTS

PARTICIPANT FLOW:
Groups:
- AKL-T03: Tablet-based game aimed at improving processing speed and attention.
- AKL-T09: Control, tablet-based word-finding game
Period: Overall Study
Arm/Group | AKL-T03 | AKL-T09
Started | 23 | 21
Completed | 20 | 20
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- AKL-T09: Control, tablet-based word finding game
- Total: Total of all reporting groups
Arm/Group | AKL-T03 | AKL-T09 | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 37
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (14.0) | 49.2 (10.9) | 51.1 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 17 | 18 | 35
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Change in Processing Speed After 6 Weeks of Treatment With a Digital Therapeutic 'Game 1', vs. 'Game 2'.
Description: Processing speed is being measured by the Symbol Digit Modalities Test (SDMT) score. SDMT measures the time to pair abstract symbols with specific numbers. The test requires visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items in 90 seconds. (max=110, min=0). Higher scores indicate improvement. Lower scores indicate worsening.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T03 | AKL-T09
Number analyzed (Participants) | 20 | 20
score on a scale | 6.10 (4.62) | 3.55 (7.51)

2. Secondary Outcome: Number of Participants With at Least 4-point Increase in SDMT Above Their Baseline Value 8 Weeks After Treatment
Description: Number of participants showing a clinically meaningful 4+ point increase in SDMT (symbol digit modalities test) relative to baseline SDMT score. Comparison of SDMT changes 8 weeks after end of treatment with Tool 1 vs. Tool 2.
Time Frame: 14 weeks
Population: 39 participants (97.5%) returned for Visit 3
Measure: Count of Participants; unit: Participants
Arm/Group | AKL-T03 | AKL-T09
Number analyzed (Participants) | 20 | 19
Participants | 14 | 7

3. Other Pre Specified Outcome: Change in Mood After 6 Weeks Treatment With Game 1 vs. Game 2
Description: Comparison of changes in mood (depression, anxiety). Depression measured using the Center for Epidemiologic Studies Depression Scale (CES-D). Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology. Anxiety measured using the State-Trait Anxiety Inventory - State subtest (STAI-S) and the State-Trait Anxiety Inventory - Trait subtest (STAI-T). Both have 20 questions and a score range 20-80, with higher scores indicating greater anxiety.
Time Frame: Baseline and 6 weeks
Population: Missing data for 6 participants on trait anxiety (STAI-T), 3 per study group; as well as for 2 participants on depression (CES-D) and state anxiety (STAI-S) measures, 1 per study group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T03 | AKL-T09
Number analyzed (Participants) | 19 | 19
score on a scale
  Depression (CES-D) | 1.11 (6.14) | -.90 (5.57)
  Anxiety - State (STAI-S) | .05 (4.64) | .21 (8.93)
  Anxiety - Trait (STAI-T): number analyzed (Participants) | 17 | 17
  Anxiety - Trait (STAI-T) | .77 (4.10) | .35 (3.35)

4. Other Pre Specified Outcome: Change in Fatigue After 6 Weeks Treatment With Game 1 vs. Game 2.
Description: Fatigue is being measured by the Modified Fatigue Impact Scale (MFIS) which has participants rank 21 items on 1 to 4 (never to always) scale. The score is the sum of these subscales. (max=84, min=0) Lower scores indicate improvement. Higher scores indicate worsening.
Time Frame: Baseline and 6 weeks
Population: Missing fatigue survey data (MFIS) for 2 participants, 1 per study group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T03 | AKL-T09
Number analyzed (Participants) | 19 | 19
score on a scale | -4.79 (6.27) | -2.95 (9.55)

5. Other Pre Specified Outcome: Change in a Digital Cognitive Battery After 6 Weeks Treatment With Game 1 vs. Game 2.
Description: Comparison of changes in scores on Match, a tablet-based assessment of processing speed and executive function. Performance is gauged on a continuous scale using the total number of correct responses given in 2-minutes. The minimum possible score is 0 (no correct responses) with higher scores indicating better performance (no maximum possible score).
Time Frame: Baseline and 6 weeks
Population: Match data was unavailable for some participants (n = 6, 3 per group)
Measure: Mean (Standard Deviation); unit: number of correct responses
Arm/Group | AKL-T03 | AKL-T09
Number analyzed (Participants) | 17 | 17
number of correct responses | 0.94 (3.54) | 0.35 (4.66)

6. Other Pre Specified Outcome: Change in Paper and Pencil Cognitive Testing After 6 Weeks Treatment With Game 1 vs. Game 2.
Description: Comparison of changes in cognition, as assessed using the BICAMS battery (Brief International Cognitive Assessment for Multiple Sclerosis) and PASAT (Paced Auditory Serial Addition Test). The BICAMS battery is composed of 3 tests (for all, higher scores indicate better performance): (1) The Symbol Digit Modalities Test (SDMT), a measure of information processing speed where performance is gauged by the number of correct responses given in 90-seconds, with a minimum possible score of 0 and maximum of 110. (2) The California Verbal Learning Test-II (CVLT-II) is a 5-trial auditory/verbal learning test with a total min. score of 0 and max of 80. (3) The Brief Visuospatial Memory Test -- Revised (BVMT-R) is a visual and spatial memory test given in 3 trials with a total min score of 0 and max of 36.
  The PASAT is a test of information processing and attention with a minimum score of 0 and maximum of 60. Higher scores indicate better performance.
Time Frame: Baseline and 6 weeks
Population: Missing PASAT data for 3 participants, 2 in AKL-T03 and 1 in AKL-T09. Data for other measures (SDMT, BVMT-R and CVLT-II) were collected from all participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKL-T03 | AKL-T09
Number analyzed (Participants) | 20 | 20
score on a scale
  SDMT | 6.10 (4.62) | 3.55 (7.51)
  CVLT-II | 2.05 (9.14) | 5.20 (8.60)
  BVMT-R | 0.70 (4.47) | 3.25 (5.23)
  PASAT: number analyzed (Participants) | 18 | 19
  PASAT | 2.72 (5.41) | 2.53 (7.19)

ADVERSE EVENTS:
Time Frame: Duration of the 6-week intervention period between Visits 1 and 2
Arm/Group | AKL-T03 | AKL-T09
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03569618/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT03569618/SAP_001.pdf